CLINICAL TRIAL: NCT05766358
Title: Role Of Metabolic Adaptation In Weight Regain: Expend Follow-Up
Brief Title: Role Of Metabolic Adaptation In Weight Regain
Acronym: EXPEND-FU
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Eric Ravussin, Associate Executive Director for Clinical Science, Pennington Biomedical Research Center
Other Study IDs: PBRC 2022-027
Record Dates: First submitted 2023-02-21; First posted 2023-03-13 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Weight Loss; Weight Gain; Obesity
MeSH Terms: conditions — Weight Loss; Weight Gain; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Placebo
  Interventions: Behavioral: Intensive lifestyle change therapy
- Tirzepatide
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Behavioral: Intensive lifestyle change therapy — Participant of both groups will be followed for 24 months after completing the parent trial intervention, with no intervention during the follow-up
  Groups: Placebo
Drug: Tirzepatide — Participant of both groups will be followed for 24 months after completing the parent trial intervention, with no intervention during the follow-up
  Groups: Tirzepatide

SUMMARY:
In a previous study (NCT04081337), 55 participants with obesity participated on a 18-week lifestyle intervention to reduce their body weight, targeting 10% body weight loss. The participants received tirzepatide (15mg after titration) or placebo during the weight loss intervention. Before and after the lifestyle intervention, energy expenditure (48-h room indirect calorimetry) and body weight and composition (dual-X-ray absorptiometry) were measured, thus enabling the assessment of metabolic adaptation. In this study, participants having provided their consent to be re-contacted will be invited to attend the research center 12,18 and 24 months after completing the lifestyle intervention. Body weight and composition will be measured, aiming to explore the association between metabolic adaptation and changes in body weight and composition after a weight loss intervention. In addition, we will explore whether weight and fat mass changes are different between groups, and whether these effects are mediated by metabolic adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Having participated in the study NCT04081337.

Exclusion Criteria:

* Being pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants having completed the NCT04081337 study.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Body weight | 24 months

SECONDARY OUTCOMES:
Body weight | 12 months
Body weight | 18 months
Body fat mass (DXA) | 12 months
Body fat mass (DXA) | 18 months
Body fat mass (DXA) | 24 months
Body fat free mass (DXA) | 12 months
Body fat free mass (DXA) | 18 months
Body fat free mass (DXA) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States